CLINICAL TRIAL: NCT01592981
Title: Subcutaneous Bortezomib, Cyclophosphamide and Rituximab (BCR) Versus Fludarabine, Cyclophosphamide and Rituximab (FCR) for Initial Therapy of Waldenstrőm's Macroglobulinaemia (WM): a Randomized Phase II Trial
Brief Title: Randomised Trial in Waldenstrom's Macroglobulinaemia
Acronym: R2W
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/11/0353
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Waldenstrom's Macroglobulinaemia
Keywords: Waldenstrom's macroglobulinaemia; bortezomib; cyclophosphamide; rituximab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Cyclophosphamide; Rituximab; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bortezomib, cyclophosphamide, rituximab (Experimental): Bortezomib:1.6 mg/m2 s.c; days 1, 8, 15 of each cycle. Cyclophosphamide:250 mg/m2 oral; days 1, 8, 15 of each cycle. Rituximab: 375 mg/m2 i.v. infusion; days 1, 8, 15 and 22 of cycles 2 and 5 only.
  Cycle repeated every 28 days. After 3 cycles of treatment, patients are reassessed and those with evidence of progression stop trial treatment. All other patients continue with further 3 cycles (to a total of 6) unless a clear clinical contradiction to further treatment exist.
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Biological: Rituximab
- fludarabine, cyclophosphamide, rituximab (Active Comparator): Fludarabine:40 mg/sq m, oral, days 1,2 and 3 of each cycle. Cyclophosphamide:250 mg/sq m; oral, days 1, 2 and 3 of each cycle. Rituximab: 375 mg/sq m i.v. infusion days 1, 8, 15 and 22 of cycles 2 and 5 only.
  Cycle repeated every 28 days.After 3 cycles of treatment, patients are reassessed and those with evidence of progression stop trial treatment. All other patients continue with further 3 cycles (to a total of 6) unless a clear clinical contradiction to further treatment exist.
  Interventions: Drug: Cyclophosphamide; Biological: Rituximab; Drug: Fludarabine

INTERVENTIONS:
Drug: Bortezomib — 1.6 mg/m2 subcutaneous bortezomib on days1, 8 and 15 of 28 days cycle
  Other Names: Velcade
  Arms: bortezomib, cyclophosphamide, rituximab
Drug: Cyclophosphamide — Cyclophosphamide:250 mg/sq m, oral, days 1, 8 and 15 of each cycle in the experimental arm.
  Cyclophosphamide:250 mg/sq m, oral, days 1, 2 and 3 of each cycle in the control arm.
Biological: Rituximab — Rituximab: 375 mg/m2 i.v. infusion; days 1, 8, 15 and 22 of cycles 2 and 5 only
  Other Names: MabThera
Drug: Fludarabine — Fludarabine: 40 mg/sq m, oral, days 1, 2 and 3
  Arms: fludarabine, cyclophosphamide, rituximab

SUMMARY:
The purpose of this trial is to assess tolerability and efficacy of the Bortezomib, Cyclophosphamide and Rituximab combination as initial therapy for previously untreated patients with symptomatic Waldenstrom's macroglobulinaemia.

DETAILED DESCRIPTION:
Waldenstrom macroglobulinaemia (WM) is a low grade nonHodgkin lymphoma characterised by bone marrow infiltration and the presence of an abnormal protein in the blood (IgM paraprotein. Most patients require treatment at presentation but there is no agreed standard of first line therapy. Current treatment is unsatisfactory with responses often incomplete and slow to attain, while recurrence is inevitable.

The aim of this study is to find out whether a new combination of Bortezomib (Velcade®), Cyclophosphamide and Rituximab (MabThera), is well tolerated and effective for patients with WM. R2W is a randomised, noncomparative, phase II trial of subcutaneous bortezomib, cyclophosphamide, rituximab (BCR, experimental arm) versus fludarabine, cyclophosphamide, rituximab (FCR, control arm) for initial therapy of WM. This is a two stage trial where six patients will be treated initially with BCR to assess tolerability. If BCR is considered tolerable, a further 50 patients will be randomised between BCR and FCR (2:1) in the second stage of the trial. Patients will receive 3 cycles of treatment and then be reassessed. Those with evidence of progression will stop trial treatment. All other patients will continue with a further 3 cycles (to a total of 6) unless there is a clear clinical contraindication to further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of WM (according to consensus panel / WHO criteria) with measurable IgM paraprotein
* Previously untreated disease at any stage requiring therapy at the discretion of the treating physician. Suggested criteria for initiating treatment include:

  * haematological suppression to Hb <10 g/dl, or neutrophils <1.5x109/l or platelets <150x109/l
  * clinical evidence of hyperviscosity
  * bulky lymphadenopathy and/or bulky splenomegaly
  * presence of B symptoms
* No previous chemotherapy (prior plasma exchange and steroids are permissible)
* Performance status grade 0 - 2
* Life expectancy of greater than 6 months
* Informed consent
* Agreed compliance with recommended contraceptive precautions where appropriate

Exclusion Criteria:

* Lymphoplasmacytic lymphoma with no detectable serum IgM paraprotein
* Severe pre-existing neuropathy (> grade 2)
* Autoimmune cytopenias
* Evidence of active Hepatitis B or C infection (patients with evidence of past HepB infection may be eligible - see appendix 6)
* Serological positivity for HIV
* Pregnant or lactating women
* Life expectancy severely limited by other illness
* Renal failure (creatinine clearance <30 ml/min)
* Severe impairment of liver function: alkaline phosphatase/bilirubin >2.5 times upper limit of normal (ULN), ALT/AST >2.5 times ULN not related to lymphoma (patients with Gilbert syndrome are eligible)
* History of allergic reaction to compounds containing boron or mannitol
* Known hypersensitivity to murine compounds.
* Diagnosed or treated for a malignancy other than WM within 5 years before day 1 of Cycle 1 with the exception of complete resection of basal cell carcinoma, squamous cell carcinoma of the skin or any other in situ malignancy
* Active systemic infection requiring treatment
* Concurrent treatment with another investigational agent
* Severe or life-threatening cardiac, pulmonary, neurological, psychiatric or metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03 (Actual); Study Completion 2020-08-02 (Actual)

PRIMARY OUTCOMES:
Disease response | 6 months (end of treatment)
  Number and percentage of patients who achieve disease response

SECONDARY OUTCOMES:
Toxicity of grade 3 or higher adverse event | Up to 6 months after treatment start
  The number and percentage of patients who experience grade 3 or higher adverse event
Progression free survival | up to 5 years after treatment start
  Time from date of randomisation to the date of first progression, relapse or death from any cause
Overall survival | up to 5 years after treatment start
  Time form date of randomisation to the date of death from any cause
Quality of life (EQ-5D score) | at 3 and 6 months after treatment start
  Quality of life will be measured using patient-completed EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Auer, Principal Investigator — St. Bartholomew's Hospital
Locations (30):
- United Kingdom (30):
  - Basingstoke & North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Birmingham Heartlands Hospital, Birmingham
  - City Hospital, Birmingham
  - Pilgrim Hospital, Boston
  - Colchester General Hospital, Colchester
  - Darent Valley Hospital, Dartford
  - Dewsbury and District Hospital, Dewsbury
  - Royal Devon and Exeter Hospital, Exeter
  - Grantham and District Hospital, Grantham
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - St Bartolomew's Hospital, London
  - University College Hospital, London
  - King's College Hospital, London
  - Northwick Park Hospital, London
  - Royal Free Hospital, London
  - Maidstone Hospital, Maidstone
  - Derriford Hospital, Plymouth
  - Pontefract Hospital, Pontefract
  - Queen's Hospital, Romford
  - Tunbridge Wells Hospital, Royal Tunbridge Wells
  - Salisbury District Hospital, Salisbury
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay
  - Pinderfields Hospital, Wakefield
  - Sandwell Hospital, West Bromwich
  - Royal Hampshire County Hospital, Winchester